CLINICAL TRIAL: NCT05995912
Title: Efficacy and Safety of Etoricoxib-tramadol 120mg/100mg on Acute Pain After Impacted Lower Third Molar Extraction: A Double Blind Randomized Controlled Trial
Brief Title: Efficacy and Safety of Etoricoxib-tramadol Tablet in Acute Postoperative Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Liomont (Industry)
Collaborators: Infinite Clinical Research, S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LT-04-20; LT-04-20 (Other: COFEPRIS, Mexico)
Record Dates: First submitted 2023-08-01; First posted 2023-08-16 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Acute Pain; Postoperative Pain
Keywords: Etoricoxib-tramadol; Third molar extraction; Analgesia
MeSH Terms: conditions — Acute Pain; Pain, Postoperative; Agnosia | interventions — Naproxen; Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etoricoxib-Tramadol (Experimental): Etoricoxib-Tramadol 120mg/100mg tablet, once-daily, for 3 days
  Interventions: Drug: etoricoxib-tramadol
- Naproxen + Tramadol (Active Comparator): Naproxen 220 mg tablet + Tramadol 50 mg capsule, twice a day, for 3 days.
  Interventions: Drug: Naproxen; Drug: Tramadol

INTERVENTIONS:
Drug: etoricoxib-tramadol — Oral administration (with or without food)
  Arms: Etoricoxib-Tramadol
Drug: Naproxen — Oral administration (with or without food)
  Arms: Naproxen + Tramadol
Drug: Tramadol — Oral administration (with or without food)
  Arms: Naproxen + Tramadol

SUMMARY:
The goal of the present phase IIb clinical trial was to compare the safety and efficacy of the fixed-dose combination etoricoxib-tramadol 120mg/100mg tablet (once a day, for three days) versus naproxen 220mg tablet plus tramadol 50 mg capsule in patients with acute postoperative pain after impacted third molar extraction. The main research question was: Is the analgesic efficacy of etoricoxib-tramadol 120mg/100mg tablet non-inferior to naproxen 220 mg tablet + tramadol 50 mg capsule in a clinical model of moderate to severe acute pain? After informed consent, patients were randomly assigned to one of the two arms: test product (etoricoxib-tramadol 120mg/100mg tablet) or active comparator (naproxen 220mg tablet + tramadol 50 mg capsule). After surgery, patients were requested to start the treatment with study drugs (test product was administered once daily for three days; meanwhile reference drug was administered twice a day for three days).

Investigators compared the effects of both treatments on pain intensity at different time frames using the visual analogue scale. Furthermore, the safety of investigational drugs was assessed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged from 18 to 40 years.
* Patients who agreed to participate in the study by signing the informed consent.
* Patients with indication for surgical extraction of impacted lower third molars according to the Pell and Gregory classification.
* Healthy subjects or with history of controlled chronic non-communicable diseases or that can be controlled prior to surgery, which, in the investigator's opinion, do not represent an additional risk for the patient.
* Patients who, at the investigator's discretion, meet personal and family conditions that allow them to properly comply with the activities described in the protocol and adherence to treatment.

Exclusion Criteria:

* Findings in the clinical history, vital signs, physical examination or laboratory studies suggesting abnormal conditions which represent a risk for subject's health at the investigator´s discretion.
* Hypersensitivity to any of the active ingredients and/or excipients of the investigational drugs.
* Patients with active peptic or gastroduodenal ulcer or diagnosis 30 days prior to signing the informed consent.
* Patients with history of allergic asthma reactions.
* Patients with severe hepatic dysfunction, classified as Child Pugh C or when being less, the investigator considers it an additional risk for patients.
* Patients with a creatinine clearance <30 mL/min.
* Patients with coagulation disorders.
* Patients with Systemic Lupus Erythematosus.
* Patients with congestive heart failure (NYHA class II-IV), ischemic heart disease, peripheral arterial disease, or cerebrovascular disease who have recently (3 months) undergone coronary artery bypass grafting or angioplasty procedures.
* Patients at high risk of acute cardiovascular events (intense smoking, hypertension or uncontrolled diabetes mellitus).
* Patients with a history of systemic neoplastic diseases or under treatment with chemotherapy.
* Patients with a history of illicit drug abuse or addiction to alcohol or tobacco.
* Patients with monoamine oxidase inhibitors (MAOIs) treatment or during the last 2 weeks prior to the study drug administration.
* Patients with opioid analgesics, neuromodulators, or long-acting NSAIDs therapy who, according to medical criteria, cannot carry out a withdrawal scheme for at least five half-lives prior to surgery.
* Patients with history of seizures or who are under treatment with medications that reduce the seizure threshold and who, according to medical criteria, cannot carry out a withdrawal scheme within 30 days prior to surgery.
* Positive pregnancy test or lactating women.
* Positive rapid urine drug test.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
Pain intensity difference (PID) | At 4 h (Day 0, postdosing) respect the baseline (Day 0, before dosing)
  The difference in pain intensity at 4 h after drug administration versus time 0 (baseline, before dosing)

SECONDARY OUTCOMES:
Pain intensity difference (PID) | At 1, 2, 3, 6, 12, 24, 48, and 72 hours postdosing respecto the baseline (Day 0, before dosing)
  The difference in pain intensity at 1, 2, 3, 6, 12, 24, 48, and 72 hours after drug administration versus time 0 (baseline, before dosing)
Total pain relief (TOTPAR) | At 4, 6, 12, 24, 48, 72 hours postdosing respect to the baseline (Day 0, before dosing)
  TOTPAR is a time-weighted measure of AUC or total area under the pain relief curve and is a summary measure that integrates serial assessments of a subject's pain over the duration of the study or in any time frime.
Trismus control | At the end of the study (Day 7) respect to the baseline (Day 0, before dosing)
  Measurement the difference of mouth opening (in mm) at baseline (before dosing) and at the end of the study (Day 7).
Adverse events | From informed consent (Day -28) to the end of the study (Day 7)
  Characteristics and frequency of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Tania A. Sibaja Ponce, M.D., Principal Investigator — Oaxaca Site Management Organization, S.C.
Locations (1):
- Oaxaca Site Management Organization, Oaxaca City, Mexico

IPD SHARING:
Plan to Share IPD: No